CLINICAL TRIAL: NCT00157742
Title: An Open Single-Centre Parallel Randomised Trial of Spinal Cord Stimulation (SCS) and Percutaneous Myocardial Revascularisation (PMR) in Patients With Refractory Angina Pectoris
Brief Title: Comparison of SCS and PMR in Patients With Refractory Angina Pectoris
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPIRIT
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2005-09

CONDITIONS: Angina Pectoris
Keywords: Angina Pectoris; Spinal Cord Stimulation (SCS); Percutaneous Myocardial Revascularisation (PMR); Refractory Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Spinal Cord Stimulation

INTERVENTIONS:
Procedure: Spinal Cord Stimulation (SCS)
Procedure: Percutaneous Myocardial Laser Revascularisation (PMR)

SUMMARY:
Randomised trial of Spinal Cord Stimulation (SCS) and Percutaneous Myocardial Laser Revascularisation (PMR) in patients with Refractory Angina Pectoris.

Hypothesis: difference in exercise tolerance at 12 months between SCS and PMR

DETAILED DESCRIPTION:
The purpose of this open, parallel, single-center prospective, randomised controlled trial is to compare two treatments: Spinal Cord Stimulation (SCS) and Percutaneous Myocardial Laser Revascularisation (PMR) and assess their use and longer term effect in patients with Refractory Angina Pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Patient limiting angina (CCS III or IV) despite maximally tolerated medical therapy
* Documented coronary artery disease (within the last 9 months prior baseline), which is unsuitable for conventional revascularisation techniques
* Patient has documented reversible ischemia on nuclear scan (Tc-99 sestamibi)
* Patient is limited in daily activities, primarily exercice capability, by their angina pain
* Age 18 or older
* Patient must understand the therapy and give informed consent
* Patient must be available for appropriate follow-up times for length of Study
* Non pregnant woman

Exclusion criteria:

* Not candidate for surgical implantation of SCS and/or not for PMR and/or unable to use SCS device appropriately for treatment
* Patient who has had one or more major cardiac events within 2 months
* Patient with myocardial wall thickness< 8 mm in the ischaemic area to be treated as verified by echocardiography
* Patient with extensive peripheral vascular disease that precludes vascular access required for PMR
* Patient on intravenous therapy to control their symptoms
* Patient who is unlikely to survive for more than 12 months due to non cardiac condition e.g.malignancy
* patient who has other diseases that are considered of greater clinical significance than the angina pectoris that would impact the ability of the clinician to adequately assess the incremental effects of the trial treatment
* Patient with ejection fraction of less than 30 % as verified by echocardiography
* Patient with cause of angina other than coronary artery disease (e.g. syndrome "X" patient)
* Patient who are unable to perform treadmill exercice test per protocol
* Patient who was previously enrolled in this study, or is currently in another clinical study, which will interfere with this protocol
* Patient who has has SCS , a TMLR or PMR procedure in the past
* Patient with an implanted pacemaker or defibrillator
* Patient who has medical conditions which may require Magnetic resonance Imaging (MRI)
* Patient with history of dementia or other persisting mental disorders significantly interfering with ability to cooperate or comply with the requirements of the study or comprehend informed consent
* Patient with history of Alcohol og Drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2000-09; Study Completion 2007-01

PRIMARY OUTCOMES:
Improvement in total exercice time following SCS compared to PMR at 12 months

SECONDARY OUTCOMES:
Angina measured by the CCS class and the patients subjectives observations
Morbidity/Mortality
Quality of life
Medication consumption
Difference in myocardial perfusion scanning
Myocardial ischemia during exercise treadmill testing
Safety profiles

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schofield, MD, Principal Investigator — Papworth Hospital, NHS
Locations (1):
- Papworth Hospital, Papworth Everard, Cambridge, United Kingdom